CLINICAL TRIAL: NCT05151042
Title: Digitally Fabricated Inter-occlusal Wafer Versus Wafer-less Distal Segment Repositioning for Bilateral Sagittal Split Osteotomy in Skeletal Mandibular Deformities (Randomized Controlled Trial)
Brief Title: Digital Occlusal Wafer Versus Waferless Distal Segment Repositioning for BSSO in Skeletal Mandibular Deformities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham O. Morsi, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS 3 - 3 - 7
Record Dates: First submitted 2021-10-23; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Maxillofacial Abnormalities; Jaw Abnormalities; Prognathism; Retrognathia; Micrognathism; Dentofacial Deformities; Congenital Abnormalities; Craniofacial Abnormalities
Keywords: Orthognathic Surgery; Orthognathic Surgical Procedures; Mandibular Advancement; Osteotomy, Sagittal Split Ramus; Mandibular Osteotomy; Computer-aided Design; 3D printing; Computer guided surgery; splint-less; computer-aided surgical simulation; virtual Mock-up surgery; Custom plate; 3D planning; Surgical guide; Osteotomy guide; repositioning guide; computer-assisted orthognathic surgery; virtual planning accuracy
MeSH Terms: conditions — Maxillofacial Abnormalities; Jaw Abnormalities; Prognathism; Retrognathia; Micrognathism; Dentofacial Deformities; Congenital Abnormalities; Craniofacial Abnormalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): Distal segments repositioning using osteotomy/plate locating bone-borne surgical guide (wafer-less approach).
  Interventions: Procedure: wafer-less approach
- Group II (Active Comparator): Distal segments repositioning using preoperative and final wafers.
  Interventions: Procedure: Computer Guided orthognathic surgery using occlusal wafers

INTERVENTIONS:
Procedure: wafer-less approach — Using the software, 3D digitized bony mandible will be virtually osteotomized and repositioned to the new postoperative position. CAD/CAM generated preoperative wafer will be placed on the lower arch dentition, the guide has an extension to guide medial, vertical, oblique cuts as well as screw holes for reference landmarks for proximal segment & tooth bearing segment. Drilling of all the reference landmarks on the proximal segment and locating medial, vertical, oblique cuts.
  Removal of guide, then BSSO is performed. The final wafer is placed, the guiding hole on the proximal segment will then be realigned with the previously drilled screw holes, fixation using mono cortical screws then drilling screw holes for plate fixation.
  Fixation of the osteotomy using 2.0 mm pre-bent mini plates.
  Arms: Group I
Procedure: Computer Guided orthognathic surgery using occlusal wafers — Using the software, 3D digitized bony mandible will be virtually osteotomized and repositioned to the new postoperative position.
  dental casts will be scanned dental casts are superimposed to the CT cuts into the virtual software environment to produce final wafer CAD/CAM repositioning guide. the generated preoperative wafer will be placed on the lower arch dentition, the guide has an extension to guide medial, vertical, oblique cuts as well as screw holes for reference landmarks for proximal segment & tooth bearing segment.
  Drilling of all the reference landmarks on the proximal segment and locating medial, vertical, oblique cuts. Removal of guide, then BSSO is performed.
  The final wafer is placed, the guiding hole on the proximal segment will then be realigned with the previously drilled screw holes, fixation using mono cortical screws then drilling screw holes for plate fixation.
  Fixation of the osteotomy using 2.0 mm pre-bent mini plates.
  Arms: Group II

SUMMARY:
Research studies continues to attempt testing modifications to refine the treatment protocols through computer assisted design or computer-generated surgical Wafer splints, have greatly revolutionized the incorporation of digital imaging and 3D design in Orthognathic surgery.

Integrating computer guided technology in orthognathic surgery aims to to simplify workup and reduce surgical errors, eliminate occlusal discrepancy, increase the realignment accuracy of the distal segments according to the preoperative plan. Implementing a waferless technique raised the question of efficiency versus the use of occlusal wafers and whether it has a significant measurable effect on the surgical outcome and objectives.

Rationale for conducting this study is to assess the difference between the effect of computer guided waferless technique and computer guided technique with occlusal wafer on accuracy of postoperative occlusion and condylar position.

.

DETAILED DESCRIPTION:
The use of waferless orthognathic surgery technique raised the question of efficiency versus the use of occlusal wafers and whether it has a significant measurable effect on the surgical outcome and objectives.

Modification and attempts to refine the treatment protocols through computer assisted design or computer-generated surgical Wafer splints, have greatly revolutionized the incorporation of digital imaging and 3D design in Orthognathic surgery. Combining the knowledge acquired from later studies with the advancement in 3D design software and increased resolution of imaging, waferless orthognathic computer guided protocols have been explored and investigating a more accurate technique is now being competitively pursued. The objective of this study is to evaluate the accuracy of the 3D printed positioning device to reposition the Distal segments according to the preoperative virtual plan after BSSO versus final digitally fabricated interocclusal wafer with distal extension for correction of class II or III mandibular deformities.

Trial design:

Randomized controlled trial

From the selected eligible patient population, candidates will be randomly allocated into 2 groups:

Group I (Interventions assessment group):

Distal segments repositioning using osteotomy/plate locating bone-borne surgical guide (wafer-less approach).

Group II (Comparator group):

Distal segments repositioning using preoperative and final wafers.

Preoperative measures:

A thorough preoperative assessment of all patients carried out including history taking, clinical, photographic, and radiographic examinations in addition to dental casts analysis.

Preoperative radiographic examination:

A panoramic radiography will be requested from all patients for preliminary survey to rule out the presence of any intra-bony pathologic lesions that may interfere with surgery. Preoperative Computed Tomography (CT) of the head and neck region will be acquired for all patients utilizing multi-slice CT machine according to the following protocol:

1. Axial slices thickness: 1 mm thick or thinner.
2. Distance between slices: 1 mm or less.
3. Gantry should not be tilted (gantry tilt = 0).
4. 2D axial images in DICOM format will recorded in the CD.
5. FOV should be limited, but all the region of interest described in the request should be included. The patient's mouth should be kept open during CT scanning to ensure the separation between mandible and maxilla.
6. Voxel ratio should be 1:1 (pitch = 1:1).
7. The window should be standard, in the original format of the CT scanner.

Group I:

Work Up and Plan Execution

1. Virtual planning: Using the software, 3D digitized bony mandible will be virtually osteotomized and repositioned to the new postoperative position.
2. Printing of corrected 3D mandibular model and plate pre-bending:

   2.0 titanium mini plates will be selected and perfectly adapted over the printed corrected 3D mandibular model, as all cases will be prepared.
3. Scanning of plate adapted on the corrected model:

   Pre-bent plates will be scanned using optical scanner to generate virtual model.
4. Construction of cutting/screw hole locating guide:

Using the 3D modelling software computer guiding device will be designed to fit on Bony surfaces, osteotomy cutting guide, distal segment repositioning guide according to the 3D virtual plan with hubs fitting the 2.0 mini plates, that were previously scanned and will be used to fix the segments in place.

Surgical Procedures:

1. Owbgeser incision will be performed to expose the buccal and lingual aspects of the ramus angle region.
2. CAD/CAM generated guide will be placed on bony surfaces of the mandibles with an extension to guide medial, vertical, oblique cuts as well as screw holes for reference landmarks for proximal and distal segments.
3. Drilling of all the reference screw holes on the proximal and distal segments and locate medial, vertical, oblique cuts.
4. Removal of the guide, then BSSO is performed
5. Fixation of the osteotomy using 2.0 mm pre-bent mini plates.
6. Debridement, irrigation of the surgical field followed by wound closure and suturing.

Group II:

Work Up and Plan Execution:

1. Virtual planning: Using the software, 3D digitized bony mandible will be virtually osteotomized and repositioned to the new postoperative position.
2. Construction of preoperative and final wafers with distal extension: Patients' dental casts will be scanned and digitized into a virtual 3D model and superimposed to the CT cuts into the virtual plan software environment in order to produce final wafer CAD/CAM repositioning guide.

Surgical Procedures:

1. Owbgeser incision will be performed to expose the buccal and lingual aspects of the ramus angle region.
2. CAD/CAM generated preoperative wafer will be placed on the lower arch dentition, the guide has an extension to guide medial, vertical, oblique cuts as well as screw holes for reference landmarks for proximal segment & tooth bearing segment.
3. Drilling of all the reference landmarks on the proximal segment and locating medial, vertical, oblique cuts.
4. Removal of guide, then BSSO is performed
5. The final wafer is placed, the guiding hole on the proximal segment will then be realigned with the previously drilled screw holes, fixation using mono cortical screws then drilling screw holes for plate fixation.
6. Fixation of the osteotomy using 2.0 mm pre-bent mini plates.

Strategies to improve adherence to intervention protocol:

Face-to-Face adherence reminder session will take place in the initial visit. This session will include informing the patient about the study steps and maintain oral hygiene.

Subsequent sessions will occur at the follow-up visits. Participants will be asked about any problems they are having like pain, swelling and oral hygiene.

Patients will be recalled for clinical evaluation every week for one month and three months postoperative.

Post-operative care:

Postoperative instructions:

1. Cold compresses in the form of ice packs will be applied for 20 minutes every hour for the first 24 hours postoperatively to minimize edema.
2. All patients will be kept on the following regimen until they are discharged from the hospital.
3. Ampicillin/sulbactams1 1500 mg vial IM injection every 12 hours for 5 days.
4. Oral Metronidazole2 500 mg every 8 hours for 5 days
5. Diclofenacpotassuim3 50 mg tablets will be given every 8 hours for control of pain.
6. Diclofenac sodium4 75 mg IM injection whenever needed.
7. Dexamethasone sodium phosphate5 8 mg IM injection on 8 doses, the first 4 doses will be given every 6 hours, and then it will be tapered on next 4 doses to half the dose every 6 hours.
8. Methylprednisolone acetate6 80 mg IM injection will be given with the last dose of Epidrone.
9. The oral antibiotic regimen (Amoxicillin/Clavulanic acid 1000 mg every 12 hours)7 will be continued for 5-7 days postoperatively to guard against infection.

Postoperative assessment and follow up: All patients will be advised to stay on a soft diet for 4-6 weeks to avoid any undue forces on the surgical site.

Postoperative CT will be obtained, immediately postoperative and 6 months later respectively (intervals T3 and T4).

14.Participant timeline: Patient will be treated in 3 visits Visit Time Procedure Visit 1 (T1) Week 1 Primary diagnosis, primary impression, consent signing and preoperative radiograph (CT) with stent Visit 2 (T2) Week 2 Surgical procedure. Visit 3 (T3) Week 3 Clinical assessment & postoperative CT Visit 4 (T4) Week 27 Follow up assessment.

Sample size:

This study will be conducted for 24 patients.

Recruitment:

Patients seeking treatment at the outpatient clinic of Oral and Maxillofacial Surgery department- Cairo University will be screened for participating in the project, until the target population is reached.

Data collection, management, and analysis:

Data collection methods:

Plans to promote participant retention & complete follow-up:

* The patient's ID number, full name, telephone numbers (home, mobile and work) and address (home and work) will be recorded to be used if needed.
* Reminder phone calls will be used prior to any appointments. Plans for assessment and collection of outcomes will be at postoperative follow-up visits and through analyzing data from CTs by specialized software.

Data management:

Each patient will have a box containing all paper based and electronic data (Digital radiographic CDs, signed consent form and paper with all the data concerned with the patient and surgeries).

Statistical methods:

Categorical data will be presented as frequencies (n) and percentages (%) and will be analyzed using chi square test. Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values, and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data is normally distributed, it will be analyzed using paired t-test. If it is nonparametric, it will be analyzed using Wilcoxon signed rank test. The significance level will be set at P ≤0.05 for all tests. Statistical analysis will be performed with IBM® SPSS® Statistics Version 25 for Windows.

Monitoring 20.Data monitoring: Data will be collected by primary investigator and revised by co-supervisors and an unbiased third party.

Harms:

1. Bad split of the mandible due to several factors including the presence of impacted lower third molar, different variations of mandibular morphology, extreme of age of patients, which may cause injury inferior alveolar nerve.
2. Injury facial artery: due to improper surgical procedures.
3. Postoperative infection: due to improper postoperative care & improper usage of antibiotics, smoking, medically comprised patients with poor wound healing.
4. Bilateral mental nerve transection.
5. Infection of grafted bone.
6. Bone graft donor site infection.
7. Wound dehiscence.
8. Chronic Osteomyelitis.

Auditing:

Auditing of the study will be done by Dr .GB the main supervisor

Ethics and dissemination:

Research ethics approval: Ethical approval of such protocol will be held by Ethics Committee of Scientific Research - Faculty of Oral and Dental Medicine - Cairo University.

Protocol amendments: If any amendment is needed for the patient's greater interest and would affect the study will be discussed and approved/rejected by the Council of the department of Oral and Maxillofacial surgery, Faculty of Oral and Dental Medicine, Cairo University Informed consent: After discussing the treatment plan with the patient and educating the patient with all the data needed and complications that could be met, an Arabic consent form will be signed by the willing participants.

Confidentiality: Boxes holding all patient information will be placed in areas with limited access. Coding and numbering of the patients will be used on data collection and administrative files so not to use names and personal data on the records used.

Declaration of interest: The study is self-funded & there is no conflict of interest to declare.

Access to data: Data access is given to the principle investigators according to their needs and blinding system.

Post-trial care: Patient follow-up will continue until complete healing and therapy success

Dissemination policy: The current study results are part of the requirements for PhD degree in Oral and Maxillofacial Surgery and will be published accordingly.

All topics will be discussed by authors for future presentation and publication of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of bilateral sagittal split osteotomy for mandibular repositioning.
* All patients are free from any systemic disease that may affect normal bone healing.
* Sufficient dentition to reproduce the occlusal relationships
* Patient's consent to participate

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing
* Intra-bony lesions or infections that may interfere with surgery.
* Previous orthognathic surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Postop occlusal translational discrepancy (T3): | Outcomes will be assessed with immediate postoperative CT at T3 (week 3).
  measured in mm from sagittal, axial, and coronal postop CT images. Measuring error and deviation of postoperative bony segments to the preoperative virtual plan.
Postop occlusal translational discrepancy (T6): | Outcomes will be assessed with immediate postoperative CT at T4 (week 27).
  measured in mm from sagittal, axial, and coronal postop CT images. Measuring error and deviation of postoperative bony segments to the preoperative virtual plan.
Postop occlusion rotation and deviation (T3): | Outcomes will be assessed with immediate postoperative CT at T3 (week 3).
  measured in degrees from 3D objects preoperative 3D cephalometric landmarks. comparing postoperative occlusal plane rotational deviation in reference to preoperative planned occlusion.
Postop occlusion rotation and deviation (T27): | Outcomes will be assessed with immediate postoperative CT at T4 (week 27).
  measured in degrees from 3D objects preoperative 3D cephalometric landmarks. comparing postoperative occlusal plane rotational deviation in reference to preoperative planned occlusion.
3D spatial deviation error (T3): | Outcomes will be assessed with immediate postoperative CT at T3 (week 3).
  Absolute point to point 3D measurements in the 3D virtual environment of the postop 3D bony segments in reference to the preop objects.
3D spatial deviation error (T27): | Outcomes will be assessed with immediate postoperative CT at T4 (week 27).
  Absolute point to point 3D measurements in the 3D virtual environment of the postop 3D bony segments in reference to the preop objects.

SECONDARY OUTCOMES:
Relapse over time: | at week 27, after 6 weeks
  The aggregate of the primary outcomes time frame into error and deviation over time to show amount of the repositioned bony segments using the interventional waferless treatment protocol versus the control group using the condylar positioning arms connected to the occlusal wafers.
Operative Time | immediate postop.
  measuring the operative time of the orthognathic surgical procedure, from first incision to closure between the interventional waferless approach and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Omara, PhD, Study Chair — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Cairo University; Hesham O Morsi, MDSc, Principal Investigator — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Cairo University
Locations (1):
- Mohamed Omara, Cairo, El-Manial, Egypt